CLINICAL TRIAL: NCT02768844
Title: Physiology and Therapeutic Management of Neonatal Abstinence Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H00006578
Record Dates: First submitted 2016-05-02; First posted 2016-05-11 (Estimated); Last update posted 2025-03-20 (Actual); Status verified 2020-12

CONDITIONS: Neonatal Abstinence Syndrome
Keywords: Stochastic Resonance; Fetus/Newborn Infant; Drug Withdrawal; Substance Abuse
MeSH Terms: conditions — Neonatal Abstinence Syndrome; Substance Withdrawal Syndrome; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- SVS vs Control (Experimental): Prospective, within-subject design. Compare effects of mattress SVS (ON) and Control (SVS OFF) on physiology in opioid-exposed newborns. SVS is alternated in intervals between continuous stimulation (ON) and no stimulation (OFF/Control) throughout inter-feed intervals. The order of the ON-OFF cycles is randomized across subjects and counterbalanced between feeding periods within subjects.
  Interventions: Device: Stochastic Vibrotactile Stimulation (SVS); Other: Control

INTERVENTIONS:
Device: Stochastic Vibrotactile Stimulation (SVS) — The infant's isolette mattress will be replaced with a specially designed mattress (non-commercially available; designed by Wyss Institute, Harvard University, Cofab Design LLC) to provide gentle vibrations and sounds during mattress stimulations.
Other: Control — Absence of mattress Stochastic Vibratory Stimulation (SVS)

SUMMARY:
The overall purpose of this project is to to quantify the physiology of neonatal drug withdrawal and develop non-pharmacological techniques to help improve the therapeutic management of Neonatal Abstinence Syndrome (NAS).

DETAILED DESCRIPTION:
Novel approaches to diagnosing and treating Neonatal Abstinence Syndrome (NAS) are needed for reducing prolonged pharmacological management, minimizing hospitalization and improving developmental outcomes in drug exposed newborns. This study seeks to examine the physiology and symptoms of drug withdrawal (e.g., irritability marked by movement activity; cardio-respiratory instabilities) in infants exposed to drugs in utero and test whether sensory stimuli (tactile, auditory) reduce dysregulated systems in the withdrawing infant.

Candidates at-risk for NAS due to fetal drug exposure will be identified to investigators by the infant's primary medical caregiver. Investigators will use a modified-consecutive sampling technique, restricted by equipment and personnel availability, for enrolling infants. Participants will be studied throughout their hospitalization. Effects of stimulation will be examined at different stages of withdrawal. Efficacy of stimulation will be examined as a potential complementary treatment of NAS.

ELIGIBILITY:
Inclusion Criteria:

Eligible subjects are infants currently inpatient in the NICU or Newborn Nursery at University of Massachusetts Memorial Hospital and:

* Full-term infants (>37 wks gestational age) and late preterm infants (34-37 wks gestational age)
* Newborns at risk for NAS due to fetal-drug exposure
* At-risk infants will be infants who present with confirmed meconium and/or urine toxicology report (documented in medical chart review) for opioids (e.g., methadone, buprenorphine/subutex, oxycodone, heroin); may also have prenatal exposure to benzodiazepines, barbiturates, amphetamines, cannabinoids, alcohol, nicotine and/or caffeine.

Exclusion Criteria:

Eligible infants meeting the inclusion criteria above will be excluded from participation in the study if he/she:

* Born less than <34 weeks.
* Has a congenital abnormality
* Has a fetal anomaly
* Has hydrocephalus or intraventricular hemorrhage >grade 2
* Has a seizure disorder not related to drug withdrawal
* Has a clinically significant shunt
* Requires mechanical respiratory support

Ages: 1 Day to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 46 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2014-01-23 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
Change in Infant Movement between Mattress ON and Mattress OFF (control) | Single sessions throughout course of hospitalization. Each session may last up to 24 hours.
  Measure mean change in infant movement activity via limb sensors
Change in Infant Breathing between Mattress ON and Mattress OFF (control) | Single sessions throughout course of hospitalization. Each session may last up to 24 hours.
  Measure mean change in infant respiratory rate via respiratory inductance plethysmography (RIP)
Change in Infant Heart Rate between Mattress ON and Mattress OFF(control) | Single sessions throughout course of hospitalization. Each session may last up to 24 hours.
  Measure mean change in infant heart rate via Electrocardiography (ECG).

SECONDARY OUTCOMES:
Change in Infant Temperature between Mattress ON and Mattress OFF (control) | Single session throughout course of hospitalization. Each session may last up to 24 hours.
  Measure mean change in axillary temperature via temperature sensor.

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth B Salisbury, Ph.D., Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- University of Massachusetts Medical School, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bloch-Salisbury E, Rodriguez N, Bruch T, McKenna L, Goldschmidt L. Physiologic dysregulation in newborns with prenatal opioid exposure: Cardiac, respiratory and movement activity. Neurotoxicol Teratol. 2022 Jul-Aug;92:107105. doi: 10.1016/j.ntt.2022.107105. Epub 2022 May 27. PMID 35636580
- [Derived] Pahl A, Young L, Buus-Frank ME, Marcellus L, Soll R. Non-pharmacological care for opioid withdrawal in newborns. Cochrane Database Syst Rev. 2020 Dec 21;12(12):CD013217. doi: 10.1002/14651858.CD013217.pub2. PMID 33348423